CLINICAL TRIAL: NCT04263649
Title: Prospective Observational Study of the Power PICC Family of Devices and Accessories
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-19PICCEU01
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Peripherally Inserted Central Catheter
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All subjects: patients who require a PICC
  Interventions: Device: Peripherally Inserted Central Catheter

INTERVENTIONS:
Device: Peripherally Inserted Central Catheter — insertion of a Peripherally Inserted Central Catheter (PICC)

SUMMARY:
Post-market, observational study to collect prospective data related to the safety and performance of the Power PICC family of devices and its accessories in a real-world setting.

DETAILED DESCRIPTION:
Single-arm, post-market, observational, prospective study to asses the safety and performance of the Power PICC Power PICC family of devices and its accessories in a real-world setting. The study will only enroll patients that need a Power PICC catheter as part of their medical care. Patients will be followed from insertion through removal, or up to 180 days (whichever comes first). Data collected will be gathered from the patient's medical chart.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, regardless of age or gender, for which the investigator has decided that one of the PowerPICC study devices for either short-or long-term venous access should be inserted as standard of care
* Expected to be available for observation through the duration of PICC therapy (including outpatient therapy, if applicable)
* Provision of signed and dated informed consent form (Note: Consent of guardian or parent may be required for patients under the age of 18 years; participant assent may be required as well.)

Exclusion Criteria:

* Presence of any device-related infection, bacteremia, or septicemia is known or suspected
* Body size is insufficient to accommodate the size of implanted device
* Known or suspected to be allergic to materials contained in the device
* History of irradiation of prospective insertion site
* Previous episode(s) of venous thrombosis or vascular surgical procedures at the prospective placement site
* Local tissue factors which would prevent proper device stabilization and/or access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients who require a PICC device in a primary care facility.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Hoerauf, MD, Study Director — Becton, Dickinson and Company
Locations (14):
- Austria (2):
  - Klinikum Klagenfurt, Klagenfurt
  - Medizinische Universität Wien, Vienna
- University Hospitals KU Leuven, Leuven, Belgium
- Fakultní nemocnice Olomouc, Olomouc, Czechia
- Sygehus Soenderjylland, Sønderborg, Sønderborg, Denmark
- Universitätsklinikum Jena, Jena, Germany
- Italy (5):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont
  - Ospedale Civile di Ivrea, Ivrea, Piedmont
  - A.O.U Città della Salute e della Scienza Torino, Ospedale Molinette, Turin, Piedmont
  - Ospedale Centrale di Bolzano, Bolzano, Trentino-Alto Adige
  - Azienda Ospedaliera dei Colli - Monaldi, Napoli
- HAGA Ziekenhuis, The Hague, Netherlands
- Hospital Universitari de Girona Dr Josep Trueta, Girona, Spain
- Institut für Diagnostische und Interventionelle Radiologie, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Troubil M, Capozzoli G, Mussa B, Hodne M, Hoerauf K, Alsbrooks K. Performance and safety of PowerPICC catheters and accessories: a prospective observational study. BMJ Open. 2024 Sep 30;14(9):e081288. doi: 10.1136/bmjopen-2023-081288. PMID 39349374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centers in 9 European countries. The first participant was enrolled on June 18, 2020 and the last participant had the last study visit on January 05, 2022.
  The choice of the specific device type, size, number of lumens, and length required for an individual patient was left to the discretion of the clinician.
Pre-assignment Details: In this post market study, 450 patients, who were to receive a PICC from the PowerPICC family as per routine clinical practice, were observed for up to 180 days after device's insertion or until removal of the device because the therapy was completed, changed or cancelled. Patients, who died during the study and had the device in place at the time of death, were considered as having completed the therapy.
Groups:
- All Subjects: Patients who received a device from the BD PowerPICC family according to the clinical practice.
Period: Overall Study
Arm/Group | All Subjects
Started (A total of 451 patients signed the ICF. As 1 patient was a screening failure, the study device was attempted to be placed in 450 patients (safety set). The study device could not be placed in 2 patients and in 1 patient the study device was placed but could not be used for the intended treatment. Hence, 447 patients received treatment via the study device (evaluable set).) | 450
Receive Treatment Via the Study Device | 447
Completed (In the end of eCRF study form, 335 patients were documented as having completed the therapy via study device (device either removed because therapy was completed, changed, or cancelled or still in place at 180 days) and 115 patients were documented as non-completed.) | 335
Not Completed | 115
Not completed — Adverse Event | 53
Not completed — Lost to Follow-up | 3
Not completed — Death | 29
Not completed — Device deficiency | 19
Not completed — other reasons | 11

BASELINE CHARACTERISTICS:
Population: Patients who underwent placement of a study device.
Arm/Group | All Subjects
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] — The patients' age ranged from 6 to 96 years with a median age of 62.0 years.
  years | 60 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 439
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 40
  Austria | 16
  Belgium | 10
  Czechia | 59
  Denmark | 59
  Italy | 212
  Switzerland | 27
  Germany | 21
  Spain | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 26.30 (5.27)
Relevant medical history [Count of Participants; unit: Participants]
  Implantable devices | 11
  Past and/or current anatomical abnormalities of the central venous system | 6
  Past and/or current atrial fibrillation or other atrial arrhythmias that affects the p-wave | 36
  Known absence of a p-wave | 6
  Abnormalities of the arms | 7
  Abnormalities of the chest wall | 5
  History of coagulopathy | 9
  History of hypercoagulopathy | 2
  Current treatment with anticoagulants | 27
  Central venous access devices | 93
  History of LN dissection/ lymphedema | 49
  Renal impairment | 4
  History of phlebitis | 7
  History of venous thrombosis | 13
  History of deep vein thrombosis | 10
  History of catheter related bloodstream inf. | 4
  Other relevant medical history | 161
Primary diagnosis for current admission [Count of Participants; unit: Participants]
  Cardiac | 12
  Trauma | 2
  Neurological | 8
  Infection | 42
  Surgical | 29
  Oncological | 328
  Vascular | 4
  Gastrointestinal | 18
  Other | 7
Reason for PICC placement [Number; unit: participants] — A subject may report more than 1 reason for PICC placement.
  participants
    Central venous pressure monitoring | 2
    Hydration support | 20
    Intravenous therapy: immunoglobulins | 2
    Intravenous therapy:antimicrobial/antifungal | 79
    Intravenous therapy:blood product and transfusion | 21
    Intravenous therapy: chemotherapy | 313
    Intravenous therapy:pain management | 30
    Intravenous therapy: total parenteral nutrition | 50
    Intravenous therapy: vasopressors | 4
    Limited peripheral access | 125
    Nutritional support | 15
    Other includes post covid pancreatytis therapy and hypertension IV pharmacotherapy | 3
    Serial blood sampling | 61
    Serial radiographic studies | 3
    Thrombocytopenia or coagulopathy | 3
Intended access duration [Count of Participants; unit: Participants]
  Long-term (>=30 days) | 353
  Short-term (<30 days) | 97
Catheter insertion - Location of procedure performance [Count of Participants; unit: Participants]
  Bedside | 190
  Interventional radiology | 108
  Other | 152
Catheter insertion - Catheter tip repositioning [Count of Participants; unit: Participants]
  Catheter tip not repositioned | 19
  Catheter tip repositioned | 430
  Missing information - no study device placed | 1
Catheter insertion - Device placement successful [Count of Participants; unit: Participants]
  Device placement successful | 448
  Device placement unsuccessful | 2
Catheter insertion - Placement of catheter [Count of Participants; unit: Participants]
  Right arm | 257
  Left arm | 193
Catheter insertion - Vein accessed [Count of Participants; unit: Participants]
  Basilic | 253
  Cephalic | 15
  Brachial | 180
  Other | 2
Catheter insertion - Vessel/catheter ratio done prior to insertion [Count of Participants; unit: Participants]
  Vessel/catheter ratio done prior to insertion | 272
  Vessel/catheter ratio not done prior to insertion | 178
Catheter insertion - Number of insertion attempts [Count of Participants; unit: Participants]
  Number of insertion attempts=1 | 408
  Number of insertion attempts=2 | 32
  Number of insertion attempts=3 | 8
  Number of insertion attempts=4 | 1
  Number of insertion attempts=5 | 1
Catheter insertion - Local anesthesia used [Count of Participants; unit: Participants]
  Local anesthesia used | 448
  Local anesthesia not used | 2
Catheter insertion - Catheter length trimmed [Count of Participants; unit: Participants]
  Catheter length trimmed | 300
  Catheter length not trimmed | 150
Catheter insertion - Tunneling used [Count of Participants; unit: Participants]
  Tunneling used | 26
  Tunneling not used | 424
Catheter insertion - Sherlock TLS used [Count of Participants; unit: Participants]
  Sherlock TLS used | 0
  Sherlock TLS not used | 450
Catheter insertion - Sherlock 3CG used [Count of Participants; unit: Participants]
  Sherlock 3CG used | 259
  Sherlock 3CG not used | 191
Catheter insertion - Method to confirm catheter tip positioning [Count of Participants; unit: Participants]
  X-ray | 157
  Sherlock 3CG | 202
  Other | 91
Catheter insertion - Stabilization method [Count of Participants; unit: Participants]
  StatLock | 390
  SecurAcath | 59
  Missing information - no study device placed | 1
Catheter insertion - Dressing type [Count of Participants; unit: Participants]
  Transparent semi-permeable membrane | 410
  Gauze | 10
  Other | 29
  Missing information - no study device placed | 1
Catheter insertion - PICC insertion as per Instructions For Use (IFUs) [Count of Participants; unit: Participants]
  PICC inserted as per the IFUs | 449
  Missing information - no study device placed | 1
Catheter insertion - presence of a second implanted line vascular access device [Count of Participants; unit: Participants]
  Presence of a second implanted line vascular access device | 90
  No presence of a second implanted line vascular access device | 360

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: Incidence of Symptomatic Venous Thrombosis in Patients With a Device From the BD PowerPICC Family Used for Both Short- and Long-term Venous Access.
Description: Incidence of symptomatic venous thrombosis defined as any new occurrence of symptomatic venous thrombosis defined by thrombus presence by ultrasonography or other imaging.
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: Since the study device could not be placed in 2 patients and in 1 patient the study device was placed but could not be used for the intended treatment, these 3 subjects were excluded from the denominator for safety variable. Therefore, 447 out of 450 subjects have been considered for denominator calculation.
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Groups:
- All Subjects: Patients who require the insertion of a device from the BD PowerPICC family according to the clinical practice.
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 1.6 [0.6 to 3.2]

2. Primary Outcome: Primary Performance: Percent of PICCs That Remain in Place Through the Required Therapy Time Period.
Description: PICCs remaining in place through the required therapy time period were defined as PICCs that were either still in place at the end of the 180-day observation or had been removed because the therapy was completed (end of useful medical use), changed or cancelled. Most patients who died during the study had the device still in place at the time of death and hence were considered as having completed the therapy.
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: A total of 447 patients received treatment via the study device and were included in the evaluable set, used for the primary performance calculation.
  The percentage of PICCs that remains in place through the completion of therapy (success) was calculated by dividing successful cases by the total number of devices with non-missing data on success/failure.Therefore, 2 subjects lost to follow-up were not included in the calculation of percentage.
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 445
% of subjects after PICC placement | 81.8 [77.9 to 85.3]

3. Secondary Outcome: Secondary Safety: Incidence of Phlebitis
Description: Incidence of phlebitis where phlebitis is defined inflammation of the cannulated vessel identified by redness, swelling, warmth, tenderness, and/or cord formation
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 0 [0.0 to 0.8]

4. Secondary Outcome: Secondary Safety: Incidence of Extravasation
Description: Incidence of extravasation where extravasation is defined as accidental infiltration of a vesicant or chemotherapeutic drug into the tissue around the catheter
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 0 [0.0 to 0.8]

5. Secondary Outcome: Secondary Safety: Incidence of Local Infection
Description: Incidence of any new occurrence of local infection
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 4.5 [2.8 to 6.8]

6. Secondary Outcome: Secondary Safety: Incidence of Local Infection as Presence of Pus at the Exit Site and/or Culture Confirmed Site Infection
Description: Incidence of local infection where local infection is defined as presence of pus at the exit site and/or culture confirmed site infection
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 3.1 [2.8 to 6.8]

7. Secondary Outcome: Secondary Safety: Incidence of Catheter-related Bloodstream Infection.
Description: Incidence of Catheter-related bloodstream infection where Catheter-related bloodstream infection is defined as positive blood culture(s) with a microorganism not related to another source (e.g., UTI) OR positive blood culture(s) with microorganism matching catheter tip culture OR blood cultures from peripheral venous puncture and PICC positive with the same microorganism.
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 1.6 [0.6 to 3.2]

8. Secondary Outcome: Secondary Safety: Incidence of Accidental Dislodgement.
Description: Incidence of Accidental dislodgement where Accidental dislodgement is defined as catheter accidentally dislodged the extent to which it requires replacement.
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 447
% of subjects after PICC placement | 3.8 [2.2 to 6.6]

9. Secondary Outcome: Secondary Safety: Incidence of Vessel Laceration.
Description: Incidence of vessel laceration where vessel laceration is defined as a tear in the tissue of the vessel.
Time Frame: from insertion though removal or 180 days, whichever comes first
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 450
% of subjects after PICC placement | 0.4 [0.1 to 1.6]

10. Secondary Outcome: Secondary Safety: Incidence of Vessel Perforation.
Description: Incidence of vessel perforation where vessel perforation is defined as a hole formed in the vessel.
Time Frame: from insertion though removal or 180 days, whichever comes first
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 450
% of subjects after PICC placement | 0.2 [0.0 to 1.2]

11. Secondary Outcome: Secondary Performance: Percent of Patent Catheters
Description: Percent of patent catheters defined as the number of functional catheters through therapy/total number of catheters.
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: A total of 447 subjects received treatment via the study device and were included in the evaluable set, used for the performance calculation. However, 2 subjects were lost to follow-up and were not included in the calculation of percentage.
  Patent catheters are defined as functional catheters through therapy.
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 445
% of subjects after PICC placement | 93.9 [91.3 to 96.0]

12. Secondary Outcome: Secondary Performance: Percent of Placement Success in Single Insertion Attempt
Description: Percent of placement success in single insertion attempt defined as placement success defined as single insertion attempt, proper tip location, and patent catheter
Time Frame: during the insertion procedure
Measure: Number (95% Confidence Interval); unit: % of subjects after PICC placement
Arm/Group | All Subjects
Number analyzed (Participants) | 450
% of subjects after PICC placement | 90.4 [87.3 to 93.0]

13. Secondary Outcome: Secondary Performance - Usability: Ease of Insertion
Description: Ease of insertion determined by composite score of guidewire/stylet performance based on post-insertion survey (5 point Likert scale)
Time Frame: during the insertion procedure
Population: The analysis is based on the investigators who completed the questionnaire and answer the respective question.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 449
Participants
  Guidewire usage was easy or very easy | 419
  Force to advance the guidewire acceptable | 448
  Guidewire withdrawal/removal was easy or very easy | 425
  Force to withdraw/remove the guidewire acceptable | 448
  Guidewire integrity | 448
  Investigators were agree or strongly agree with "Guidewire facilitated placement" | 425
  Stylet usage was easy or very easy | 335
  Force to advance the stylet acceptable | 352
  Stylet withdrawal/removal was easy or very easy | 343
  Force to withdraw/remove the stylet acceptable | 353
  Stylet integrity | 356
  Investigators were agree or strongly agree with "Stylet facilitated placement" | 338

14. Other Pre Specified Outcome: Usability: Ease of Insertion When the Sherlock 3CG Pre-Loaded Stylet Used
Description: The percentage of Sherlock 3CG Pre-Loaded Stylet that aided in guidance and placement of the catheter, when used
Time Frame: during the insertion procedure
Population: The analysis is based on the investigators who completed the questionnaire and answer the respective question.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 259
Participants | 244

15. Post Hoc Outcome: Post-hoc Analysis: Device Lifetime
Description: Post-hoc analysis: overall mean device lifetime
Time Frame: from insertion though removal or 180 days, whichever comes first
Population: The overall mean device lifetime
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Subjects
Number analyzed (Participants) | 450
days | 90.64 (68.41)

ADVERSE EVENTS:
Time Frame: From PICC insertion though removal or 180 days, whichever comes first
Description: An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
  An adverse device effect is defined as any adverse event that is considered to be related to the use of an investigational medical device.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 32/450
Serious Adverse Events (participants affected / at risk) | 58/450
Other Adverse Events (participants affected / at risk) | 162/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=450)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 4 (4)
Catheter bacteraemia (Infections and infestations) | 3 (3)
Catheter site infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Germ cell cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=450)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Catheter site discharge (General disorders) | 5 (5)
Catheter site dryness (General disorders) | 2 (2)
Catheter site erythema (General disorders) | 24 (26)
Catheter site exfoliation (General disorders) | 1 (1)
Catheter site granuloma (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 3 (3)
Catheter site haemorrhage (General disorders) | 8 (8)
Catheter site hypersensitivity (General disorders) | 1 (1)
Catheter site irritation (General disorders) | 2 (2)
Catheter site necrosis (General disorders) | 1 (1)
Catheter site edema (General disorders) | 1 (1)
Catheter site pain (General disorders) | 8 (9)
Catheter site pruritus (General disorders) | 2 (2)
Catheter site related reaction (General disorders) | 2 (2)
Catheter site thrombosis (General disorders) | 1 (1)
Catheter site vesicles (General disorders) | 1 (1)
Complication of device remova (General disorders) | 1 (1)
Device related thrombosis (General disorders) | 16 (16)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Sensation of foreign body (General disorders) | 1 (1)
Vessel puncture site injury (General disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 4 (4)
Catheter bacteraemia (Infections and infestations) | 7 (7)
Catheter site infection (Infections and infestations) | 18 (19)
Device related infection (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Germ cell cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
Device dislocation (Product Issues) | 17 (17)
Device occlusion (Product Issues) | 5 (7)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 17 (21)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Oesophageal operation (Surgical and medical procedures) | 1 (1)
Venous perforation (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI submits to Sponsor for review a draft 90 days prior to submission of the draft for publication.Draft shall not divulge any confidential info.Sponsor has the right to:review and make comments on any proposed publication; withhold the use of its name in connection with publication;make any results from the study known to its customers and governmental agencies prior to publication.The first publication of the study results shall be made in conjunction with the results from the other PIs.

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04263649/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT04263649/SAP_001.pdf